CLINICAL TRIAL: NCT02196519
Title: Clinical Evaluation of Cohera Sylys Surgical Sealant as an Adjunct to Standard Bowel Anastomosis Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cohera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-106-0028
Record Dates: First submitted 2014-07-17; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Stoma Reversal Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Test (Experimental): All test arm subjects received Sylys Surgical sealant around anastomotic junction after closure.
  Interventions: Device: Sylys Surgical Sealant

INTERVENTIONS:
Device: Sylys Surgical Sealant

SUMMARY:
A first in human study evaluating the safety of Sylys Surgical Sealant in protecting the anastomotic junction created during a stoma reversal procedure.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Be in good general health in the opinion of the investigator with no conditions that would significantly impact wound healing as determined by medical history and review of recent concomitant medications
* Be scheduled for an ileostomy reversal procedure
* Be willing to follow instructions for incision care
* Agree to return for all follow-up evaluations specified in this protocol
* Sign informed consent

Exclusion Criteria:

* Anesthesia risk judged to be higher than ASA2
* Have severe co-morbid conditions that pose a high risk for surgery and adequate recovery (e.g., heart disease)
* Any condition involving compromised immune system
* Any condition known to effect wound healing, such as collagen vascular disease
* Known blood clotting disorder
* Be receiving antibiotic therapy for pre-existing condition or infection
* Concurrent use of fibrin sealants or other anastomosis care devices
* Be currently taking systemic steroids or immunosuppressive agents
* Have known or suspected allergy or sensitivity to any test materials or reagents
* Be participating in any current clinical trial or have participated in any clinical trial within 30 days of enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: W Bemelman, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); E Consten, Principal Investigator — Meander Medical Center- Amersfoort